CLINICAL TRIAL: NCT01220375
Title: PAV-trial: Plerixafor and Chemotherapy With Vinorelbine for Stem Cell Mobilization in Patients With Myeloma. A Pilot Phase II Study.
Brief Title: PAV-trial: Plerixafor and Chemotherapy With Vinorelbine for Stem Cell Mobilization in Patients With Myeloma
Acronym: PAV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Prof. Thomas Pabst, Department of Medical Oncology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 236/09; 2010DR2052 (Other: Swissmedic); 10-CPRS-001 (Other: Genzyme); 1795 (Other: Inselspital)
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Myeloma
Keywords: Mobilization of autologous peripheral blood progenitor cells PBPC; Autologous stem cell mobilization; Multiple Myeloma; Plerixafor
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma | interventions — Vinorelbine; Granulocyte Colony-Stimulating Factor; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Plerixafor is a bicyclam with hematopoietic stem cell-mobilizing activity. Plerixafor blocks the binding of stromal cell-derived factor (SDF-1alpha) to the cellular receptor CXCR4, resulting in hematopoietic stem cell release from bone marrow and HSC movement into the peripheral circulation.
  Interventions: Drug: Vinorelbine, G-CSF, & Plerixafor; Drug: Vinorelbine and Plerixafor; Drug: G-CSF and Plerixafor; Drug: Vinorelbine & Plerixafor on day when CD34 count is at least 15'000 CD34+ cells/ml of peripheral blood

INTERVENTIONS:
Drug: Vinorelbine, G-CSF, & Plerixafor — Patients 1-10 receive 35 mg/m2 vinorelbine i.v. on day 1, G-CSF divided in two daily doses from day 4 until collection of stem cells, and plerixafor as an i.v. application on day 8, at 08:00 AM, in the dose of 240 microg/kg b.w. Stem cell collection is initiated 4 hours later (at 12:00 PM) at day 8, if at least 20 X 103 of CD34+ cells / ml peripheral blood are detected.
Drug: Vinorelbine and Plerixafor — Patients 11-20 receive 35 mg/m2 vinorelbine i.v. on day 1 and plerixafor as an i.v. application on day 8, at 08:00 AM, in the dose of 240 microg/kg b.w. No G-CSF will be administered. Stem cell collection is initiated 4 hours later (at 12:00 PM) at day 8, if at least 20 X 103 of CD34+ cells / ml peripheral blood are detected.
Drug: G-CSF and Plerixafor — Patients 21-30 receive G-CSF divided in two daily doses from day 4 until collection of stem cells, and plerixafor as an i.v. application on day 8, at 08:00 AM, in the dose of 240 microg/kg b.w. No chemotherapy with vinorelbine will be gine on day 1. Stem cell collection is initiated 4 hours later (at 12:00 PM) at day 8, if at least 20 X 103 of CD34+ cells / ml peripheral blood are detected.
Drug: Vinorelbine & Plerixafor on day when CD34 count is at least 15'000 CD34+ cells/ml of peripheral blood — Patients 31-40 receive 35 mg/m2 vinorelbine i.v. on day 1 and plerixafor as an i.v. application at 08:00 AM, on the first day on which the CD34 count has risen to at least 15'000 CD34+ cells/ml of peripheral blood. Stem cell collection is initiated 4 hours later (at 12:00 PM) on this day. No G-CSF will be administered.

SUMMARY:
High-dose chemotherapy with autologous stem cell support is the current standard procedure in the first-line treatment in younger patients with myeloma fit for intensive treatment. Current practice in Switzerland for stem cell mobilization is the combination of chemotherapy and G-CSF stimulation in myeloma patients fit for high-dose chemotherapy with melphalan and autologous stem cell transplant. In this trial the intravenous application of Plerixafor is being investigated in respect of the capability of the mobilization of stem cells from the bone marrow into the peripheral blood. In contrast to the twice daily application of G-CSF (eg. Neupogen) for several days, Plerixafor has to be injected just one-time.

DETAILED DESCRIPTION:
Background

High-dose chemotherapy with autologous stem cell support is the current standard procedure in the first-line treatment in younger patients with myeloma fit for intensive treatment. Current practice in Switzerland for stem cell mobilization is the combination of chemotherapy and G-CSF stimulation in myeloma patients fit for high-dose chemotherapy with melphalan and autologous stem cell transplant. For mobilization chemotherapy, a single dose of vinorelbine is commonly used, producing mild myelosuppression. G-CSF is started at day 4 on a daily basis, allowing stem cell apheresis usually at day 8. In a subsequent study, we evaluated the use of pegylated G-CSF given as a single injection at day 4 together with vinorelbine. We found this regimen equally feasible, reliable and allowing collection of stem cells in an equally high percentage. In the current proposal, we suggest to continue this line of research investigating the mobilization using chemotherapy with vinorelbine. We propose to study the feasibility of this mobilization chemotherapy in the absence of growth factors, thus without G-CSF, in combination with Plerixafor.

Objective

Primary objective: To assess the feasibility of collection of > 6 million CD34+ peripheral blood stem cells/kg body weight in 2 days.

Secondary objectives: Assessment of safety of plerixafor during mobilization and collection of peripheral blood stem cells; feasibility of intravenous plerixafor application and stem cell apheresis in a one-day procedure on an ambulatory basis; evaluation of engraftment of peripheral blood stem cells mobilized by vinorelbine and plerixafor; evaluation of the costs for mobilization with plerixafor.

Methods

Chemotherapy with vinorelbine is given at a standard dose at day 1, on an ambulatory basis.

In part A (10 patients), G-CSF is given s.c., divided in two daily doses starting at day 4 until collection of stem cells. Plerixafor is given as an i.v. application on day 8 in the dose of 240 microg/kg b.w. Stem cell collection is initiated 4 hours later at day 8, if at least 20 x 103 of CD34+ cells / ml peripheral blood are detected. In case of insufficient collection, the procedure is repeated at day 9, including repetition of plerixafor application.

Part B (30 patients): If the combination of plerixafor and vinorelbine is found feasible and in the absence of unexpected toxicity, additional 30 patients will be studied in part B of this study. No G-CSF will be administered in part B, otherwise the treatment plan is as it is in part A.

High dose Melphalan will be used as conditioning regimen. After transplantation, G-CSF will be given to subjects starting at day +5 after PBPC reinfusion.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic stage I or stage II and III myeloma patients after standard first-line non-melphalan containing induction treatment. Patients must be fit for subsequent consolidation with high-dose chemotherapy with melphalan with autologous stem cell support.
* Standard induction chemotherapy comprises regimens including thalidomide, bortezomib, or lenalidomide (up to 4 cycles), alone or in combination with dexamethasone. Combinations of novel agents are allowed as well as induction with the VAD regimen.
* Patients must have achieved at least a partial response according to the Bladé criteria after induction chemotherapy.
* Patient must be aged 18-70 years, with an ECOG < 2 and has given voluntary written informed consent.
* Platelets count 50 x 109/l without transfusion support within 7 days before the laboratory test.
* Absolute neutrophil count (ANC) 1.0 x 109/l without the use of colony stimulating factors.
* Corrected serum calcium < 3 mmol/L.
* Aspartate transaminase (AST) <= 1.5 x ULN.
* Alanine transaminase (ALT) <= 1.5 x ULN.
* Total bilirubin <= 2 x ULN.
* Creatinin-clearance >= 50 ml/min.
* Negative pregnancy test within 14 days prior to registration for all women of childbearing potential. Patients of childbearing potential must implement adequate measures to avoid pregnancy during study treatment and for additional 12 months. No pregnant or lactating patients are allowed.

Exclusion Criteria

* Patients previously treated with melphalan or extensive radiotherapy to the bone marrow.
* Patients with more than 4 cycles of chemotherapy with Lenalidomide.
* Patients not fit for autologous stem cell transplantation.
* Patient receiving colony stimulating factors.
* Patient underwent plasmaphereses within 4 weeks before enrolment.
* Patient had major surgery within 4 weeks before enrolment.
* Patient has other serious medical condition that could potentially interfere with the completion of treatment according to this protocol or that would impair tolerance to therapy or prolong hematological recovery.
* Sero-positive for HIV antibody.
* Patient known to be hepatitis B surface antigen positive or who has an active hepatitis C infection.
* Patient has an active systemic infection requiring treatment.
* Female patient is pregnant or breast feeding.
* Compromised renal function as evidenced by measured or calculated creatinine clearance <= 50 ml/min.
* Subject is currently enrolled in, or has not yet completed at least 30 days since ending another investigational device or drug trial or is receiving other investigational agent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of patients from whom ≥ 6 million CD34+ peripheral blood stem cells/kg are harvested in a maximum of 2 days | day 8 (and 9, if necessary) / 2 days after G-CSF

SECONDARY OUTCOMES:
Incidence and severity of adverse events during and after the use of plerixafor | 15 days
Proportion of patients with engraftment of PBPC defined as an ANC recovery of ≥ 0.5 x 109/L for 3 consecutive days and a platelet recovery of ≥ 20 x 109/L in the absence of platelet transfusion for at least 7 days | 21 months
Comparison of costs for mobilization of PBPC with vinorelbine and plerixafor versus the costs for mobilization with vinorelbine and filgrastim and versus the costs for mobilization with vinorelbine and pegfilgrastim | 21 Months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pabst, Associate Professor, Principal Investigator — Dep. Medical Oncology, Bern University Hospital
Locations (1):
- Dep. of Medical Oncology, Bern University Hospital, Bern, Switzerland